CLINICAL TRIAL: NCT02898714
Title: The Impact of Flash Glucose Monitoring on Clinical Outcome Parameters in Diabetes Patients
Brief Title: Flash Glucose Monitoring Study for Diabetes
Acronym: FUTURE
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof dr Pieter Gillard, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: FUTURE-59342
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
On the first of July 2016, the Freestyle Libre Flash Glucose Monitor (FGM) will be reimbursed in Belgium by means of a new diabetes reimbursement program for adults. For children, the Freestyle Libre FGM is also reimbursed by means of a new reimbursement program from the first of August 2016 onwards. Making this the only way to receive the device in Belgium. To understand the impact of this new FGM on diabetes patients in UZ Leuven, OLVZ Aalst, and UZ Antwerp, we want to study the use of the device by our patients by means of an observational study where patients complete questionnaires at regular time points in the first year of usage and after 24 months Clinical data will be gathered during the routine clinical visits as part of the reimbursement program.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* >= 4 years
* Using flash glucose monitoring

Exclusion Criteria:

* Doesn't want to sign the informed consent
* < 4 years
* Not using flash glucose monitoring

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older than 4 years with diabetes using FGM after entering in the new diabetes reimbursement program in Belgium in UZ Leuven, OLVZ Aalst and UZ Antwerp.
Sampling Method: Non-Probability Sample
Enrollment: 2331 (Actual)
Dates: Start 2016-07; Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Quality of life | 12 months
  Change in quality of life measures from baseline to 12 months

SECONDARY OUTCOMES:
Quality of life | 24 months
  Change in quality of life measures from baseline to 24 months
HbA1c | 12 months
  Change in HbA1c from baseline to 12 months
HbA1c | 24 months
  Change in HbA1c from baseline to 24 months
Severe hypoglycaemia | 12 months
  Change in severe hypoglycaemia frequency from baseline to 12 months
Severe hypoglycaemia | 24 months
  Change in severe hypoglycaemia frequency from baseline to 24 months
Time in hypoglycaemia (<54 mg/dL and <70 mg/dL) | 12 months
  Change in time spent in hypoglycaemia (<54 mg/dL and <70 mg/dL) from baseline to 12 months
Time in hypoglycaemia (<54 mg/dL and <70 mg/dL) | 24 months
  Change in time spent in hypoglycaemia (<54 mg/dL and <70 mg/dL) from baseline to 24 months
Hospitalisations because of hypoglycaemia and/or ketoacidosis | 12 months
  Change in number of hospitalisations because of hypoglycaemia and/or ketoacidosis from baseline to 12 months
Hospitalisations because of hypoglycaemia and/or ketoacidosis | 24 months
  Change in number of hospitalisations because of hypoglycaemia and/or ketoacidosis from baseline to 24 months
Work and school absenteeism | 12 months
  Change in work and school absenteeism from baseline to 12 months
Work and school absenteeism | 24 months
  Change in work and school absenteeism from baseline to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Meulemeester J, Charleer S, Visser MM, De Block C, Mathieu C, Gillard P. The association of chronic complications with time in tight range and time in range in people with type 1 diabetes: a retrospective cross-sectional real-world study. Diabetologia. 2024 Aug;67(8):1527-1535. doi: 10.1007/s00125-024-06171-y. Epub 2024 May 24. PMID 38787436
- [Derived] Charleer S, De Block C, Bolsens N, Van Huffel L, Nobels F, Mathieu C, Gillard P. Sustained Impact of Intermittently Scanned Continuous Glucose Monitoring on Treatment Satisfaction and Severe Hypoglycemia in Adults with Type 1 Diabetes (FUTURE): An Analysis in People with Normal and Impaired Awareness of Hypoglycemia. Diabetes Technol Ther. 2023 Apr;25(4):231-241. doi: 10.1089/dia.2022.0452. Epub 2023 Feb 3. PMID 36648249
- [Derived] Broos B, Charleer S, Bolsens N, Moyson C, Mathieu C, Gillard P, De Block C. Diabetes Knowledge and Metabolic Control in Type 1 Diabetes Starting With Continuous Glucose Monitoring: FUTURE-PEAK. J Clin Endocrinol Metab. 2021 Jul 13;106(8):e3037-e3048. doi: 10.1210/clinem/dgab188. PMID 33740049
- [Derived] Charleer S, De Block C, Van Huffel L, Broos B, Fieuws S, Nobels F, Mathieu C, Gillard P. Quality of Life and Glucose Control After 1 Year of Nationwide Reimbursement of Intermittently Scanned Continuous Glucose Monitoring in Adults Living With Type 1 Diabetes (FUTURE): A Prospective Observational Real-World Cohort Study. Diabetes Care. 2020 Feb;43(2):389-397. doi: 10.2337/dc19-1610. Epub 2019 Dec 16. PMID 31843948